CLINICAL TRIAL: NCT05222893
Title: Optimization of Positive End-expiratory Pressure During Laparoscopic Surgery
Brief Title: Optimization of PEEP During Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaganda Medical University (Other)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other); National Research Oncology and Transplantology Center, Kazakhstan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PEEP-TPP
Record Dates: First submitted 2021-11-24; First posted 2022-02-03 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Post-Op Complication; Ventilator-Induced Lung Injury
Keywords: positive end-expiratory pressure; esophageal pressure; laparoscopic surgery
MeSH Terms: conditions — Postoperative Complications; Ventilator-Induced Lung Injury | interventions — Capnography; Blood Gas Analysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PEEP Pes (Active Comparator): PEEP adjustment according to the pressure indicators in the lower third of the esophagus Pes (intervention group)
  Interventions: Diagnostic Test: Respiratory monitoring; Diagnostic Test: Capnography; Diagnostic Test: Arterial blood gas; Device: Esophageal pressure
- PEEP 5 (Active Comparator): PEEP constantly set at 5 cmH2O (control group)
  Interventions: Diagnostic Test: Respiratory monitoring; Diagnostic Test: Capnography; Diagnostic Test: Arterial blood gas; Device: Esophageal pressure

INTERVENTIONS:
Diagnostic Test: Respiratory monitoring — Measurement of the plateau pressure, positive end-expiratory pressure, driving pressure, end-expiratory lung volume, compliance of respiratory system on volume-controlled ventilation
Diagnostic Test: Capnography — Measurement of end-tidal carbon dioxide tension, volume of CO2 eliminated per minute
Diagnostic Test: Arterial blood gas — Measurement of the oxygen partial pressure and the carbon dioxide partial pressure
Device: Esophageal pressure — Measurement the pressure in the lower third of esophagus during inspiration and expiration

SUMMARY:
Lung-protective ventilation (LPV) during general anesthesia can trigger the development of early postoperative pulmonary complication (PPC) and ventilator associated lung injury. One of the proven components of the LPV is low tidal volume (TV). Data on the positive end-expiratory pressure (PEEP) parameters adjustment in laparoscopic surgery, as well as the effects on the respiratory biomechanics, lung tissue and respiratory muscles damage are limited and not clear.

The objective of the study is to evaluate the ability of the esophageal pressure (Pes) based controlled personalized PEEP adjustment, to improve the biomechanics of the respiratory system and oxygenation due to laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
During laparoscopic surgery pressure on alveoli increases, due to in the conditions of pneumoperitoneum, muscle relaxation, the patient's position on the operating table, excess body weight and other factors. As the consequence, the alveoli collapse due to negative transpulmonary pressure. The personalized PEEP adjustment for each particular patient during laparoscopic surgery can help to avoid the adverse effects on biomechanical parameters of the respiratory system, the early PPC incidence and improve overall patients' recovery.

The objective of the study is to evaluate the ability of the esophageal pressure (Pes) based controlled personalized PEEP adjustment, to improve the biomechanics of the respiratory system and oxygenation due to laparoscopic cholecystectomy.

Investigators will measure if PEEP adjustment according to the pressure indicators in the lower third of the esophagus Pes (intervention group) versus PEEP constantly set at 5 cmH2O (control group) gives better outcomes and prevent the early PPC incidence in hospitals.

After the induction, intubation and insertion of the esophageal balloon catheter, TV for patients both groups is set to 6 ml / kg BMI: for men (50+0.91* (height-152.4), for women (45+0.91* (height-152.4); minute ventilation (MV) to ensure the level of PetCO2 - 30-35 mmHg, respiratory rate (RR) 15-25/min (maximum up to 35/min).

Gas exchange parameters including partial pressures of oxygen (PaO2) and carbon dioxide (PaCO2) in arterial blood will be measured before the induction (T0), after 1 hour after surgery (T5) and after 24 hours after surgery (T6), then will calculate PAO2/FiO2 respectively.

FiO2, oxygen saturation (SpO2), hemodynamic parameters including blood pressure (BP), heart rate (HR) will be recorded in all point of the study.

Following respiratory mechanics will be measured: plateau pressure (Pplat), PEEP, driving pressure (DP), Pes during inspiration and expiration, volumetric capnometry (VCO2), end-tidal carbon dioxide tension (PetCO2).

Respiratory system compliance (Cstat, Cl, Ccw), end-expiratory lung volume (EELV) will calculated after intubation (T1), after PEEP set according to the patient's group allocation PEEP Pes and PEEP 5 (T2), after initiating pneumoperitoneum (T3) and placing the patient in the reverse Trendelenburg position (T4).

This is a randomized controlled study in the operating room of the University hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic surgery with mechanical lung ventilation American Society of Anesthesiologists Classification (ASA) I-III

Exclusion Criteria:

* pregnancy
* age less than 18 or more than 70 years
* patients ASA > III
* life-threatening heart rhythm abnormalities and/or systolic blood pressure < 80 mmHg despite norepinephrine at a dose > 2 μg/kg/min
* primary lung diseases (e.g. interstitial lung diseases, lung emphysema) or tumor metastases in the lungs
* chronic decompensated diseases with extrapulmonary organ dysfunction (tumor progression, liver cirrhosis, congestive heart failure)
* Glasgow coma score < 14
* upper airways obstruction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Change in arterial partial oxygen tension to inspiratory oxygen fraction (PaO2/FiO2) ratio | 5 minutes before intubation,1 hour after surgery, 24 hour after surgery
  Calculation of the arterial partial oxygen tension to inspiratory oxygen fraction (PaO2/FiO2) ratio using arterial oxygen tension measurement and compare between groups

SECONDARY OUTCOMES:
Dynamics of the end-expiratory lung volume | 5 minutes after induction and intubation, 5 minutes after PEEP setting, 5 minutes after pneumoperitoneum, 5 minutes after reverse Trendelenburg position
  Calculation the end-expiratory lung volume (ml) and compare with expected and between groups
Dynamics of the respiratory biomechanics | 5 minutes after induction and intubation, 5 minutes after PEEP setting, 5 minutes after pneumoperitoneum, 5 minutes after reverse Trendelenburg position
  Calculation the compliance of respiratory system (ml/mbar) and compare between groups at all time points
Dynamics of the volume of CO2 eliminated per minute | 5 minutes after induction and intubation, 5 minutes after PEEP setting, 5 minutes after pneumoperitoneum, 5 minutes after reverse Trendelenburg position
  Measurement of volume of CO2 eliminated per minute (VCO2 in ml/min), than compare the trends as a marker of lung ventilation
Dynamics of the partial pressure of CO2 in exhaled gas | 5 minutes after induction and intubation, 5 minutes after PEEP setting, 5 minutes after pneumoperitoneum, 5 minutes after reverse Trendelenburg position
  Measurement of partial pressure of CO2 in exhaled gas (PetCO2 in mmHg) than compare the trends as a marker of lung ventilation
Dynamics of the hemodynamic parameters | 5 minutes after induction and intubation, 5 minutes after PEEP setting, 5 minutes after pneumoperitoneum, 5 minutes after reverse Trendelenburg position
  Measurement of the arterial blood pressure (mmHg) and compare between groups at all time points

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Oncology and Transplantology Centre, Astana, Select, Kazakhstan

REFERENCES:
- [Background] Barbosa FT, Castro AA, de Sousa-Rodrigues CF. Positive end-expiratory pressure (PEEP) during anaesthesia for prevention of mortality and postoperative pulmonary complications. Cochrane Database Syst Rev. 2014 Jun 12;2014(6):CD007922. doi: 10.1002/14651858.CD007922.pub3. PMID 24919591
- [Background] Bender SP, Paganelli WC, Gerety LP, Tharp WG, Shanks AM, Housey M, Blank RS, Colquhoun DA, Fernandez-Bustamante A, Jameson LC, Kheterpal S. Intraoperative Lung-Protective Ventilation Trends and Practice Patterns: A Report from the Multicenter Perioperative Outcomes Group. Anesth Analg. 2015 Nov;121(5):1231-9. doi: 10.1213/ANE.0000000000000940. PMID 26332856
- [Background] Kacmarek RM, Villar J. Lung-protective Ventilation in the Operating Room: Individualized Positive End-expiratory Pressure Is Needed! Anesthesiology. 2018 Dec;129(6):1057-1059. doi: 10.1097/ALN.0000000000002476. No abstract available. PMID 30277931
- [Background] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507
- [Background] Iaroshetskii AI, Protsenko DN, Rezepov NA, Gel'fand BR. [Positive end-expiratory pressure adjustment in parenchimal respiratory failure: static pressure-volume loop or transpulmonary pressure?]. Anesteziol Reanimatol. 2014 Jul-Aug;59(4):53-9. Russian. PMID 25549487
- [Background] Pereira SM, Tucci MR, Morais CCA, Simoes CM, Tonelotto BFF, Pompeo MS, Kay FU, Pelosi P, Vieira JE, Amato MBP. Individual Positive End-expiratory Pressure Settings Optimize Intraoperative Mechanical Ventilation and Reduce Postoperative Atelectasis. Anesthesiology. 2018 Dec;129(6):1070-1081. doi: 10.1097/ALN.0000000000002435. PMID 30260897